CLINICAL TRIAL: NCT06352125
Title: An Observational Trial to Assess the Performance of the TEG® 6s Diagnostic System With the Citrated K, KH, RTH, FFH Cartridge
Status: Completed | Type: Observational
Sponsor: Haemonetics Corporation (Industry)
Collaborators: ClinStatDevice (Unknown); Boston Healthcare Technologies Consultants, LLC (Unknown)
Responsible Party: Sponsor
Other Study IDs: TP-CLN-100503
Record Dates: First submitted 2024-04-02; First posted 2024-04-08 (Actual); Last update posted 2024-04-08 (Actual); Status verified 2023-02

CONDITIONS: Surgery
MeSH Terms: interventions — Thrombelastography

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Whole Blood Samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

GROUPS / COHORTS (2):
- Liver Transplant
  Interventions: Diagnostic Test: TEG 6s Citrated K, KH, RTH, FFH Cartridge; Diagnostic Test: Clauss Fibrinogen
- CV Surgery
  Interventions: Diagnostic Test: TEG 6s Citrated K, KH, RTH, FFH Cartridge; Diagnostic Test: Clauss Fibrinogen

INTERVENTIONS:
Diagnostic Test: TEG 6s Citrated K, KH, RTH, FFH Cartridge — The TEG® 6s uses the Global Hemostasis with Heparin Neutralization (HN) Cartridge to test the hemostasis properties of citrated blood samples using four different assays/reagents simultaneously, one in each of the four cartridge channels.
Diagnostic Test: Clauss Fibrinogen — Diagnostic Test: Clauss Fibrinogen Fibrinogen, also known as Factor I, is a plasma protein that can be transformed by thrombin into a fibrin gel ("the clot"). Fibrinogen is synthesized in the liver and circulates in the plasma as a disulfide-bonded dimer of 3 subunit chains. The biological half-life of plasma fibrinogen is 3 to 5 days.

SUMMARY:
This clinical trial is designed to assess the agreement of the TEG® 6s system using the Citrated K, KH, RTH, FFH, cartridge (hereafter referred to as the Heparin Neutralization (HN) Cartridge) with its comparators.

ELIGIBILITY:
Inclusion Criteria:

Patients who are at an increased risk of intervention-induced coagulopathy or at increased risk of developing intervention-induced coagulopathy complications undergoing cardiovascular surgeries or liver transplantation (recipients):

1. Adult patients (18 years of age and older) who underwent cardiovascular on-pump surgeries or procedures (e.g., CABG) who were at an increased risk of coagulopathy-related complications1 (see Table 9.3-1) as well as patients with clinically apparent or suspected coagulopathy or
2. Adult patients (18 years of age and older) who underwent not-on-pump cardiovascular surgeries (e.g., lead extraction) or cardiovascular procedures (e.g., minimally invasive valve or percutaneous cardiac procedures, such as PCI, LAAC, TAVR/TAVI) associated with the use of heparin who were at an increased risk of coagulopathy-related complications1 (see Table 9.3-1) as well as patients with clinically apparent or suspected coagulopathy or
3. Adult patients (18 years of age and older) who underwent liver transplantation (recipients)

Exclusion Criteria:

1. Patients with hereditary chronic coagulation and/or bleeding disorders
2. Patients with hereditary fibrinolytic bleeding disorders
3. Patients deemed unfit for participation in the by the principal investigator
4. Patients participating in another clinical that would not be scientifically or medically compatible with this trial
5. Patients with currently altered coagulation due to the presence of oral anticoagulants (e.g., apixaban, rivaroxaban, dabigatran, warfarin)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who are at an increased risk of intervention-induced coagulopathy or at increased risk of developing intervention-induced coagulopathy complications.
Sampling Method: Non-Probability Sample
Enrollment: 338 (Actual)
Dates: Start 2021-12-09 (Actual); Primary Completion 2023-01-31 (Actual); Study Completion 2023-01-31 (Actual)

PRIMARY OUTCOMES:
Primary Method Comparison | Outcome measure from the single blood draw was assessed within 2 hours of blood draw.
  CK-MA TEG Parameter. Unit of measurement was mm.
Primary Method Comparison | Outcome measure from the single blood draw was assessed within 2 hours of blood draw.
  CKH-MA TEG Parameter. Unit of measurement was mm.
Primary Method Comparison | Outcome measure from the single blood draw was assessed within 2 hours of blood draw.
  CRTH-MA TEG Parameter. Unit of measurement was mm.
Primary Method Comparison | Outcome measure from the single blood draw was assessed within 2 hours of blood draw.
  CFFH-MA TEG Parameter. Unit of measurement was mm.
Primary Method Comparison | Outcome measure from the single blood draw was assessed within 2 hours of blood draw.
  CK-R TEG Parameter. Unit of measurement was minutes.
Primary Method Comparison | Outcome measure from the single blood draw was assessed within 2 hours of blood draw.
  CKH-R TEG Parameter. Unit of measurement was minutes.
Primary Method Comparison | Outcome measure from the single blood draw was assessed within 2 hours of blood draw.
  CKH-LY30 TEG Parameter. Unit of measurement was percentage.

CONTACTS AND LOCATIONS:
Overall Officials: Jan Hartmann, MD, Study Director — Haemonetics Corporation
Locations (7):
- United States (7):
  - University of California - San Francisco, San Francisco, California
  - University of Colorado, Aurora, Colorado
  - Ochsner Clinic, New Orleans, Louisiana
  - Lifebridge Health (Sinai Hospital), Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - University of Texas Health Science Center - San Antonio, San Antonio, Texas

REFERENCES:
- [Derived] Adelmann D, Hartmann J, Moore HB, Yockelson SR, Dageforde LA, Chitilian H, Little MB, Bliden KP, Gurbel PA, Tantry US, Subramaniam K, Sakai T. TEG (R) 6s Heparin Neutralization Cartridge for Hemostatic Assessment of Patients Undergoing Cardiovascular Surgery. Anesthesiology. 2026 Jan 1;144(1):103-115. doi: 10.1097/ALN.0000000000005759. Epub 2025 Sep 18. PMID 40965969